## Statistical plan BENEFIC STUDY

Project: Proof of Mechanism of a New Ketogenic Supplement Using Dual Tracer PET (Positron Emission

Tomography) (BENEFIC)

Clinical trial number: NCT02551419
REB reference number: MP-22-2015-509
Principal Investigator: Pr. Stephen Cunnane
Promotor: Université de Sherbrooke

Funding: Alzheimer Association US dans Nestlé Health Science

Document version: November 28, 2019

## **Description:**

6-month RCT in MCI, 2 groups (Placebo and Active), repeated measurements (2 times, PRE-POST), recruitment in two phases:

• Phase 1 (2015-2017): N=20 Placebo et N=19 Active, completed

• Phase 2 (2017-2020): n= 20 placebo and n=20 active, expected completers

• Final participant: Jan 2020

## **Statistical analysis:**

| Outcomes | Variables |
|---|---|
| Outcome I-a | Brain ketone metabolism (CMR <sub>ket</sub> and K <sub>ket</sub> ) (phase 1) |
| Outcome I-b | Blood total ketone response (phase 1 + phase 2) |
| Outcome II-a | Brain glucose metabolism (CMR <sub>glu</sub> and K <sub>glu</sub> ) (phase 1) |
| Outcome II-b | Regional CMR <sub>ket</sub> and CMR <sub>glu</sub> (phase 1) |
| Outcome II-c | Change in MRI-based parameters |
| Outcome II-d | Cognitive evaluation |
| Outcome II-e | Blood metabolite profile as a measure of safety |
| Outcome II-f | Derived Brain ketone metabolism (dCMR <sub>ket</sub> phase 2) |
| Outcome II-g | Pharmacokinetic ketone response (phase 2) |

Variables for brain energy metabolism (phase 1)

- cerebral metabolic rate of total ketones (CMR<sub>ket</sub>)
- cerebral metabolic rate of glucose (CMR<sub>glu</sub>)
- regional CMR<sub>ket</sub> and CMR<sub>glu</sub>
- Brain ketone and glucose uptake (K)

Variables for plasma ketone concentrations and derived brain ketone uptake:

- Total ketones (mM).
- Derived cerebral metabolic rate of total ketones (dCMR<sub>ket</sub>, μmol/100 g/min) (phase 2)
- Pharmacokinetic ketone response (AUC 8 hour) (phase 2)

Variables for plasma metabolites profile:

- Total cholesterol (mM).
- Triglycerides (mM).
- Glucose (mM).
- Acetoacetate (mM).
- Beta-hydroxybutyrate (mM).

Variables for cognitive evaluation:

- Raw scores for RL/RI-16, BVMT-R, Digit Symbol, Digit Span, *Trail Making Test A and B, Stroop Color and Word Tests*, *Verbal Fluency and Boston naming test*.
- Composite score for each of the five main cognitive domains (Z-score).

Variables for MRI-based parameters (phase 1)

- brain blood flow (ASL)
- brain activation (rs-fMRI)
- integrity of brain white matter tracts (dMRI)
- regional brain volumes (vMRI)

## 1) Data analysis

- Shapiro-Wilks Normality Test ->
  - o <u>parametric statistics</u> -> ANCOVA analysis With the POST measure as the dependent variable and the PRE as a covariate. This model will assess between-group differences in the POST means after accounting for PRE values (Dimitrov et Rumrill 2003). The model will also be controlled for age, education and APOE-4 genotype (if no interaction Groupe x covariable).
  - Non parametric statistics -> Intra-group PRE vs. POST (dependent samples): Wilcoxon Sign tests. Inter-group delta Placebo vs. delta Active: Mann—Whitney U tests
- Linear regression between plasma ketones and cerebral metabolic rate of total ketones (CMR<sub>ket</sub>)
- Linear regression between plasma ketones and cognitive performance.
- Linear regression between cerebral metabolic rate of total ketone (including dCMR<sub>ket</sub>) and cognitive performance